CLINICAL TRIAL: NCT03930472
Title: Testing Two Farmers Market Voucher Strategies to Increase Food Security
Brief Title: #WYMarketsMatter: Testing Two Farmers Market Voucher Strategies to Increase Food Security
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wyoming (Other)
Collaborators: Wyoming Food for Thought (Unknown)
Responsible Party: Principal Investigator, Christine Porter, Associate Professor, Wyoming Excellence Chair in Community & Public Health, University of Wyoming
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3077662143
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Food Security; Produce Consumption
Keywords: Farmers Markets; Vouchers

STUDY DESIGN:
Intervention Model Description: With delayed intervention for control group, but those outcomes not assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Voucher intervention F&V (Experimental): Receiving $20 in vouchers at each of up to 4 markets ($80 total) that are good for F&V only
  Interventions: Behavioral: Market vouchers
- Voucher intervention SNAP (Experimental): Receiving $20 vouchers at each of up to 4 markets that are good for any foods that SNAP/EBT benefits can be used for
  Interventions: Behavioral: Market vouchers
- Waitlist control (No Intervention): Delayed intervention/waitlist control (who, at the final data gathering, will receive 5 x $20 in vouchers good at the WFfT 2019 and 2020 markets).

INTERVENTIONS:
Behavioral: Market vouchers — Receiving $80 in vouchers good for fruits and vegetables or for SNAP-eligible foods at 4 out of 5 markets in late July and in August, 2019.
  Arms: Voucher intervention F&V; Voucher intervention SNAP

SUMMARY:
University of Wyoming (UW) and Wyoming Food for Thought Project (WFFTP) propose to collaboratively develop, pilot, and evaluate a trial on the impact of market vouchers on food security and fruit and vegetable (F&V) consumption. We will (a) provide farmers market vouchers to families who are enrolled in WIC, SNAP, or free or reduced lunch and/or have incomes ≤185% of poverty line; (b) assess impacts of these supports on household food security and F&V consumption; and (c) test feasibility and impacts of vouchers valid only for F&V vs. for any foods that can be purchased with SNAP.

To test the feasibility and preliminary impacts of this approach, we will enroll 30 individuals/households in this study, randomizing 10 to each of the 2 intervention arms and 10 to waitlist control. Qualifying individuals and families will be able to enroll in the study at the WFFTP Tuesday afternoon/evening market on July 30th, 2019. They will be randomized upon enrollment to one of three conditions: receiving $20 in vouchers at each of up to 4 markets ($80 total) that are good for F&V only, receiving $20 vouchers at each of up to 4 markets that are good for any foods that SNAP/EBT benefits can be used for; or delayed intervention/waitlist control (who, at the final data gathering, will receive 5 x $20 in vouchers good at the WFFTP 2019 and 2020 markets).

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the intervention, a participant must be an adult aged ≥18 years old whose household is enrolled in or eligible for SNAP, free or reduced school lunch program, and/or WIC (i.e., incomes of ≤185% of poverty for household size). UW staff wills screen for eligibility by verifying a participant has an EBT card. If no card is available, participants will be asked to self-report household income and size and UW staff will use the Federal Poverty Level chart to determine the individual's eligibility. They must also self-identify as living in Casper, Wyoming. They must come in person to the market on July 30th, 2019, to enroll.

Exclusion Criteria:

Not meeting the criteria above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Food security | five week intervention, questions for past 30 days
  USDA six-item short form Food Security Survey Module. They have been adapted to reflect food security in the previous 30 days (as opposed to 12 months) in order to compare food security before and during the intervention. Survey and tools available online at http://www.ers.usda.gov/topics/food-nutrition-assistance/food-security-in-the-us/survey-tools.aspx#.VEk0Bfl4qug
Fruit and vegetable consumption | five week intervention, questions for past 30 days
  The 16 relevant questions from the National Institutes of Health survey "Eating at America's Table Study: Quick Food Scan."

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wyoming, Laramie, Wyoming, United States

IPD SHARING:
Plan to Share IPD: No